CLINICAL TRIAL: NCT00683085
Title: Phase I/II Trial of Human Leukocyte Antigen (HLA)-A*02:01-restricted Vascular Endothelial Growth Factor Receptor 1 (VEGFR1)-Derived Peptide Vaccination Combined With Conventional Dose of Gemcitabine for Advanced Pancreatic Cancer
Brief Title: Human Leukocyte Antigen-A*02:01-restricted Tumor Vessel Specific Peptide Vaccination for Advanced Pancreatic Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of eligible patient
Sponsor: Tokyo University (Other)
Collaborators: Human Genome Center, Institute of Medical Science, University of Tokyo (Other)
Responsible Party: Naohide Yamashita MD,PhD, Research Hospital, The Institute of Medical Science, The University of Tokyo
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMSUT-PPKVEGFR10201
Record Dates: First submitted 2008-05-16; First posted 2008-05-23 (Estimated); Results first posted 2010-12-17 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Pancreatic Cancer; Pancreas Neoplasms
Keywords: cancer; pancreas; advanced; peptide; vaccination; VEGFR1; HLA; gemcitabine; IFA; Cancer of Pancreas; Neoplasms, Pancreas; Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Peptide vaccination (Experimental): VEGFR1-derived HLA-A*02:01-restricted peptide (VEGFR1-A2-770; TLFWLLLTL)was vaccinated twice weekly for 8 weeks (total 16 doses) combined with conventional dose (1,000 mg/m^2 body surface area) of gemcitabine 6 doses for advanced stage pancreatic cancer to confirm the safety and efficacy of this type of peptide.
  Interventions: Biological: HLA-A*02:01-restricted VEGFR1-derived peptide vaccination

INTERVENTIONS:
Biological: HLA-A*02:01-restricted VEGFR1-derived peptide vaccination — VEGFR1-derived HLA-A*02:01-restricted peptide (VEGFR1-A2-770; TLFWLLLTL)was vaccinated twice weekly for 8 weeks (total 16 doses) combined with conventional dose (1,000 mg/m^2 body surface area) of gemcitabine 6 doses for advanced stage pancreatic cancer to confirm the feasibility and efficacy of this type of peptide.
  Other Names: VEGFR1-A2-770; TLFWLLLTL

SUMMARY:
Pancreatic cancer is the fourth leading cause of cancer death in the United States, and no combination therapy is far superior to gemcitabine alone. Vascular endothelial growth factor receptor type 1 (VEGFR1) is expressed on the tumor vessels and a candidate of tumor vessel-specific peptide vaccination strategy to induce T cell immune response. We conducted the study to confirm the safety and efficacy of combined modality intervention using conventional dose of gemcitabine with peptide vaccination targeting tumor-vessel specific VEGFR1 in case of advanced/inoperable or therapy-resistant pancreatic cancer patients.

Gemcitabine 1,000 mg/m^2 (body surface area) will be administered on day 1, day 8, day 15, day 29, day 36, and day 43, respectively.

VEGFR1-derived HLA-A*02:01-restricted peptide (VEGFR1-A02-770; TLFWLLLTL) emulsified with Montanide ISA51 will be subcutaneously injected twice weekly for 8 weeks (total 16 doses).

DETAILED DESCRIPTION:
HLA-A*02:01-restricted VEGFR1-specific cytotoxic T lymphocyte (CTL) responses were obtained from HLA-A2/Kd transgenic murine model.

HLA-A*02:01-restricted VEGFR1-specific CTL clones were also obtained from peripheral blood mononuclear cells of healthy volunteer donors.

These CTL clones showed potent anti-tumor CTL responses in HLA class Ⅰ-restricted manner in vitro.

Vaccination of HLA-A*02:01-restricted VEGFR1-specific peptide to A2/Kd transgenic mice markedly suppress the tumor-induced angiogenesis and tumor growth in vivo.

ELIGIBILITY:
Inclusion Criteria:

* Heterozygote or homozygote of HLA-A*02:01 allele
* Inoperable or recurrent pancreatic cancer with or without any prior therapy
* Difficult to continue the prior therapy due to treatment-related toxicities
* ECOG performance status 0-2
* Evaluable primary or metastatic lesion with RECIST v.1.0 criteria
* Clearance period from prior therapy more than 4 weeks
* Life expectancy more than 3 months
* Laboratory values as follows 2,000/μL< WBC <15,000/μL Platelet count >100,000/μL AST <150 IU/L ALT <150 IU/L Total bilirubin <3.0 mg/dl Serum creatinine <3.0 mg/dl

Exclusion Criteria:

* Pregnancy (refusal or inability to use effective contraceptives)
* Breastfeeding
* Active or uncontrolled infection
* Systemic use of corticosteroids or immunosuppressants
* Uncontrollable brain metastasis and/or meningeal infiltration
* Unhealed external wound
* Possibilities of complicated paralytic ileus or interstitial pneumonitis
* Decision of not eligible determined by principal investigator or attending doctor

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2008-05; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naohide Yamashita, MD, PhD, Study Director — Director, Research Hospital, Institute of Medical Science, Tokyo University
Locations (1):
- Research Hospital, The Institute of Medical Science, The University of Tokyo, Minato-ku, Tokyo, Japan

REFERENCES:
- [Background] Nagayama H, Sato K, Morishita M, Uchimaru K, Oyaizu N, Inazawa T, Yamasaki T, Enomoto M, Nakaoka T, Nakamura T, Maekawa T, Yamamoto A, Shimada S, Saida T, Kawakami Y, Asano S, Tani K, Takahashi TA, Yamashita N. Results of a phase I clinical study using autologous tumour lysate-pulsed monocyte-derived mature dendritic cell vaccinations for stage IV malignant melanoma patients combined with low dose interleukin-2. Melanoma Res. 2003 Oct;13(5):521-30. doi: 10.1097/00008390-200310000-00011. PMID 14512794
- [Background] Ishizaki H, Tsunoda T, Wada S, Yamauchi M, Shibuya M, Tahara H. Inhibition of tumor growth with antiangiogenic cancer vaccine using epitope peptides derived from human vascular endothelial growth factor receptor 1. Clin Cancer Res. 2006 Oct 1;12(19):5841-9. doi: 10.1158/1078-0432.CCR-06-0750. PMID 17020992

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Neighboring research hospitals around Tokyo, Japan sent three candidates to our hospital during May, 2008 to March, 2009.
Pre-assignment Details: Wash out time was four weeks from preceding therapy, and three candidates were evaluated for eligibility. Two cases were compatible to our eligibility, but another candidate was excluded from this study entry because he was not expected to survive more than three months.
Groups:
- Peptide 1 mg Twice Weekly for 8 Weeks With Gemcitabine: HLA-A*0201-restricted VEGFR1-specific peptide, VEGFR1-A02-770(TLFWLLLTL) 1 mg, subcutaneous injection, twice every weeks for eight weeks (total 16 doses) combined with incomplete Freund adjuvant (IFA) and gemcitabine 1,000 mg/m^2 of body surface area
Period: Overall Study
Arm/Group | Peptide 1 mg Twice Weekly for 8 Weeks With Gemcitabine
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Peptide 1 mg Twice Weekly for 8 Weeks With Gemcitabine
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 55 (7.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Without Grade 4 Hematological or Grade 3 to 4 Non-hematological Adverse Events
Description: Number of participants without grade 4 hematological or grade 3 other adverse events were caslculated based on the National Cancer Institute Common Terminology Criteria for Adverse Events version 3.0 (NCI CTCAE v.3)
Time Frame: 2 months
Population: Intention to treat (ITT)
Measure: Number; unit: participants
Arm/Group | Peptide 1 mg Twice Weekly for 8 Weeks With Gemcitabine
Number analyzed (Participants) | 2
participants | 1

2. Secondary Outcome: Number of Participants With Tumor Regression
Description: Sum of diameters of primary pancreatic tumor or metastatic tumors (target lesions) before and after vaccination were measured by computed tomography. Sum of tumors' size diameters decrease more than 30% after vaccination was diagnosed as response according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.0 guidelines.
Time Frame: 2 months
Population: intension to treat (ITT)
Measure: Number; unit: participants
Arm/Group | Peptide 1 mg Twice Weekly for 8 Weeks With Gemcitabine
Number analyzed (Participants) | 2
participants | 0

ADVERSE EVENTS:
Time Frame: During 2 months after initiation of vaccination
Description: Serious adverse events include grade 4 hematological or grade 3 to 4 non-hematological adverse events
Arm/Group | Peptide 1 mg Twice Weekly for 8 Weeks With Gemcitabine
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peptide 1 mg Twice Weekly for 8 Weeks With Gemcitabine (N=2)
Blood in stool (Gastrointestinal disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peptide 1 mg Twice Weekly for 8 Weeks With Gemcitabine (N=2)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Leukocytes (Blood and lymphatic system disorders) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
Neutrophils (Blood and lymphatic system disorders) | 2 (2)
Platelets (Blood and lymphatic system disorders) | 1 (1)
Injection site reaction (Skin and subcutaneous tissue disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No